CLINICAL TRIAL: NCT06868914
Title: Phase I Clinical Trial to Study the Safety and After-effects of Transcranial Magnetic Stimulation (TMS) Using A High-density Theta Burst Stimulation (hdTBS) Paradigm
Brief Title: Phase I Trial of High-Density Theta Burst Stimulation (hdTBS)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 10001666; 001666-DA
Record Dates: First submitted 2025-03-10; First posted 2025-03-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Healthy Volunteers
Keywords: Substance Use Disorders (SUDs); Transcranial Magnetic Stimulation (TMS); Theta Burst Stimulation (TBS); High-density Theta Burst Stimulation (hdTBS)
MeSH Terms: conditions — Substance-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TBS (3- and 5-pulse TBS) (Active Comparator): Each participant will receive 2 active TBS (3- and 5-pulse TBS) and 1 sham TBS on 3 visits separated by at least 48 hours to minimize any potential accumulating effects from prior visits.
  Interventions: Device: TMS (MagVenture MagPro 100 with MagOption)
- Sham TBS (Sham Comparator): Each participant will receive 2 active TBS (3- and 5-pulse TBS) and 1 sham TBS on 3 visits separated by at least 48 hours to minimize any potential accumulating effects from prior visits.
  Interventions: Device: TMS (MagVenture MagPro 100 with MagOption)

INTERVENTIONS:
Device: TMS (MagVenture MagPro 100 with MagOption) — TMS will be applied using the MagVenture MagPro 100 with MagOption (MagVenture Inc, Alpharetta, GA) stimulator with a figure-of-8 TMS coil.
  Each subject will receive 2 active TBS (3- and 5-pulse TBS) and 1 sham TBS on 3 visits separated by at least 48 hours.

SUMMARY:
Background:

Transcranial magnetic stimulation (TMS) uses magnetic pulses to affect brain activity. A type of TMS called theta burst stimulation (TBS) is approved to treat people with major depression. Researchers have developed a new form of TBS called high-density TBS (hdTBS). They hope hdTBS will work better than TBS. But first they need to test the new treatment in healthy adults.

Objective:

To test hdTBS in healthy adults. Also, to compare the aftereffects of hdTBS and TBS.

Eligibility:

Healthy adults aged 22 to 60 years.

Design:

Participants will have 4 clinic visits over about 3 to 4 weeks. They must abstain from drugs and alcohol and limit caffeine before visits.

At their first visit, participants will be oriented to TBS. They will wear a cap and earplugs. A device with round coils will be placed near their head. When a brief electric current passes through the coil, it generates a magnetic pulse that stimulates the brain. Participants may feel a pulling sensation on the skin under the coil. Their fingers may move involuntarily.

At their next 3 visits, participants will receive either TBS or sham TBS. A sham TBS uses a low magnetic field to minimize the effects of the treatment. Participants will have up to 9 electrodes placed on 1 arm. These electrodes will measure the electrical activity in their muscles. Each TBS session will be videotaped.

At every visit, participants will answer questions about their health, including substance use. They will perform 2 tasks to test their thinking skills. They will perform a test on a computer to test their reaction time....

DETAILED DESCRIPTION:
Study Description:

This study is intended to test the safety and potential efficacy of the highdensity theta burst stimulation (hdTBS) paradigm. We hypothesize that hdTBS i) can be safely administered to normal healthy human subjects, and ii) can produce stronger and longer-lasting after-effects than the conventional FDA-approved TBS paradigm.

Objectives:

Primary Objective:

To determine whether hdTBS at the power level of 60% and 80% resting motor threshold can be safely administered to normal healthy human participants.

Secondary Objective:

To determine whether hdTBS produces stronger and longer-lasting after-effects than the conventional, FDA-approved TBS protocol. Here "after-effects" are defined as alterations in cortical excitability after TMS administration, which can be quantitatively assessed by measuring motor-evoked potential (MEP) before and after an acute session of TMS on the primary motor cortex. Changes in the characteristics and durations of the MEP signal relative to pre-TMS baseline reflect neuromodulation effects of the TMS session.

Endpoints:

Primary Endpoint:

Clinically significant adverse events as collected on the Noninvasive Brain Stimulation (NIBS) monitoring questionnaire and evaluated by the MAI in combination with the serious adverse event reports.

Secondary Endpoints:

20 complete datasets at the 80% RMT hdTBS dose that are evaluable for after-effects of hdTBS.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Be 22-60 years of age.

  --Justification: Many neural processes change with age, and these changes could introduce unwanted variability in behavior. In addition, the risk of difficult-to detect medical abnormalities such as silent cerebral infarcts increase with age. Children under the age of 22 are excluded from this study because safety of rTMS in children has not been studied. In addition, this study is more than minimal risk and presents no direct benefit.
* Ability and willingness to provide written informed consent.

  --Justification: Written informed consent must be obtained for this study per NIH policy and federal regulations.
* Generally in good health.

  * Justification: Many illnesses may alter neural functioning. These will be evaluated by the MAI and excluded as needed.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

-Personal history of stroke, brain lesions, previous neurosurgery, any personal history of seizure or fainting episode of unknown cause, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than two days or other neurological condition deemed by the MAI to be likely to affect response to the TBS being delivered.

* Justification: Stroke or head trauma can lower the seizure threshold, and are therefore contra indications for TMS. Fainting episodes or syncope of unknown cause could indicate an undiagnosed condition associated with seizures.

  -First-degree family history of any form of epilepsy with a potentially hereditary basis.
* Justification: First-degree family history of epilepsy with a hereditary component increases the risk of the participant having an undiagnosed condition that is associated with lowered seizure threshold.

  -Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object in the body that precludes TMS intervention.
* Justification: Any metal around the head is a contraindication for TMS, as it involves exposure to a relatively strong magnetic field.

  -Noise-induced hearing loss or tinnitus.
* Justification: individuals with noise-induced hearing problems may be particularly vulnerable to the acoustic noise generated by TMS equipment.

  -Current use (any use in the past 4 weeks, chronic use within 6 past six months) of any investigational drug or of any medications with psychotropic, anti or pro-convulsive action.
* Justification: The use of certain medications or drugs can lower seizure threshold and is therefore contraindicated for TMS.

  -Lifetime history of major depressive disorder, schizophrenia, bipolar disorder, mania, or hypomania.
* Justification: The population of interest here is a healthy control population with no psychiatric disorders. In participants with depression, bipolar disorder, mania or hypomania, there is a small chance that TMS can trigger (hypo)manic symptoms.

  -Current use of nicotine (self-report, urine cotinine test and/ or CO consistent with smoker) or history of more than 20 cigarettes or 20 instances of nicotine use in lifetime or history of daily nicotine use.
* Justification: The population of interest here is a healthy control population with no substance use disorder and therefore a minimal nicotine exposure history in the control group is required.

  -Current regular use of more than 2 cups of coffee or equivalent caffeine intake in the morning (not total daily intake).
* Justification: Excessive caffeine use can reduce seizure threshold and could potentially increase risk of TMS-induced seizure.

  -Meet current DSM-5 criteria for any substance use disorder, or urine toxicology positive for any illicit substance inconsistent with history given.
* Justification: The population of interest is a healthy control population with no substance use disorder. Current use of illicit substances could lower seizure threshold and is therefore contraindicated for TMS.

  -Have met DSM-5 criteria for any substance use disorder in the past.
* Justification: the population of interest is a healthy control population with no present or past substance use disorder.

  -History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or any heart condition currently under medical care.
* Justifications: the risk of TMS for individuals with a heart condition is unknown.

  -Pregnant individuals or individuals with reproductive potential who are sexually active and do not report using contraception.
* Justification: it is unknown whether TMS poses a risk to fetuses.

  -Otherwise TMS incompatible or have participated in any noninvasive brain stimulation (NIBS) session in the past two weeks or a NIBS treatment course in the past 6 months.
* Justification: in order to limit exposure to TMS, we will not enroll participants who have received TMS less than two weeks ago.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2028-01-13 (Estimated); Study Completion 2028-01-13 (Estimated)

PRIMARY OUTCOMES:
Clinically significant adverse events as collected on the Noninvasive Brain Stimulation (NIBS) monitoring questionnaire and evaluated by the MAI in combination with the serious adverse event reports. | about 3-4 weeks
  As a phase I trial, 25 participants are a reasonable sample size for a preliminary assessment of the safety profile of the hdTBS paradigm.

SECONDARY OUTCOMES:
20 complete datasets at the 80% RMT hdTBS dose that are evaluable for after-effects of hdTBS. | about 3-4 weeks
  20 complete datasets should give sufficient power to detect an effect. hdTBS produces stronger and longer lasting after-effects sets a solid foundation for future study in patients to investigate the efficacy of the new TMS paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Yihong Yang, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We share information with researchers outside the NIH in two ways. Most commonly, we have specific partnerships with other researchers. Also, we may put data into one or more scientific databases, where it is stored along with information from other studies. Researchers can then study the information combined from many studies to learn even more about health and disease. We will share some protocol data with our scientific research partners inside or outside the NIH. Research partners outside the NIH sign an agreement with the NIH to share data. This agreement indicates the type of data that can be shared and what can be done with those data.@@@Additionally, de-identified data may be shared with properly administered databases and/or with collaborators with whom proper data sharing agreements are in place, after consultation with and approval from the NIDA-IRP Scientific Director.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available at the time of publication and as long as the archive is online or for a minimum of 5 years after publication in the event it must be moved to new hosting archives.
Access Criteria: We may put data into one or more scientific databases, where it is stored along with information from other studies. We will share some protocol data with our scientific research partners inside or outside the NIH. Research partners outside the NIH sign an agreement with the NIH to share data. This agreement indicates the type of data that can be shared and what can be done with those data.@@@Additionally, de-identified data may be shared with properly administered databases and/or with collaborators with whom proper data sharing agreements are in place, after consultation with and approval from the NIDA-IRP Scientific Director. Data shared with NIH investigators outside of NIDA, unless otherwise stated, would be sent by NIDA as de-identified data via secure email, encryption or secured ftp. The code to those data will not be shared.